CLINICAL TRIAL: NCT03490955
Title: Effects of Black Pepper on the Absorption of Nutrients in Vegetables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-3973
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-03

CONDITIONS: Black Pepper; Absorption; Carotenoid
MeSH Terms: interventions — Condiments; Rapeseed Oil; black pepper oil; Salads; Olive Oil; Corn Oil; Sunflower Oil; Linseed Oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Salad (Sham Comparator): Subjects will consume a vegetable salad without dressing one time in the morning.
  Interventions: Other: salad
- Salad dressing (canola oil) (Active Comparator): Subjects will consume a vegetable salad with dressing (canola oil) one time in the morning
  Interventions: Other: salad dressing (canola oil)
- black pepper (Active Comparator): Subjects will consume a vegetable salad without dressing (canola oil) but with black pepper one time in the morning
  Interventions: Other: black pepper
- Salad dressing (canola oil) and black pepper (Active Comparator): Subjects will consume a vegetable salad with dressing (canola oil) and with black pepper one time in the morning
  Interventions: Other: salad dressing (canola oil) and black pepper
- Salad dressing (olive oil) and black pepper (Active Comparator): Subjects will consume a vegetable salad with dressing (olive oil) and with black pepper one time in the morning
  Interventions: Other: Salad dressing (olive oil) and black pepper
- Salad dressing (corn oil) and black pepper (Active Comparator): Subjects will consume a vegetable salad with dressing (corn oil) and with black pepper one time in the morning
  Interventions: Other: Salad dressing (corn oil) and black pepper
- Salad dressing (sunflower oil) and black pepper (Active Comparator): Subjects will consume a vegetable salad with dressing (sunflower oil) and with black pepper one time in the morning
  Interventions: Other: Salad dressing (sunflower oil) and black pepper
- Salad dressing (flaxseed oil) and black pepper (Active Comparator): Subjects will consume a vegetable salad with dressing (flaxseed oil) and with black pepper one time in the morning
  Interventions: Other: Salad dressing (flaxseed oil) and black pepper

INTERVENTIONS:
Other: salad dressing (canola oil) and black pepper — Subjects will consume a vegetable salad with black pepper and dressing (canola oil) one time in the morning
  Arms: Salad dressing (canola oil) and black pepper
Other: salad dressing (canola oil) — Subjects will consume a vegetable salad with dressing (canola oil) one time in the morning
  Arms: Salad dressing (canola oil)
Other: black pepper — Subjects will consume a vegetable salad without dressing (canola oil) but with black pepper one time in the morning
  Arms: black pepper
Other: salad — Subjects will consume a vegetable salad without dressing (canola oil) and without black pepper one time in the morning
  Arms: Salad
Other: Salad dressing (olive oil) and black pepper — Subjects will consume a vegetable salad with black pepper and dressing (olive oil) one time in the morning
  Arms: Salad dressing (olive oil) and black pepper
Other: Salad dressing (corn oil) and black pepper — Subjects will consume a vegetable salad with black pepper and dressing (corn oil) one time in the morning
  Arms: Salad dressing (corn oil) and black pepper
Other: Salad dressing (sunflower oil) and black pepper — Subjects will consume a vegetable salad with black pepper and dressing (sunflower oil) one time in the morning
  Arms: Salad dressing (sunflower oil) and black pepper
Other: Salad dressing (flaxseed oil) and black pepper — Subjects will consume a vegetable salad with black pepper and dressing (flaxseed oil) one time in the morning
  Arms: Salad dressing (flaxseed oil) and black pepper

SUMMARY:
The objective of this project is to determine the extent to which eating black pepper together with vegetables increase the absorption of carotenoids (a class of important nutrients) in the vegetables such as beta-carotene.

DETAILED DESCRIPTION:
Black pepper has multiple health-promoting effects, many of which are associated with the relatively high levels of piperine it contains. Piperine can enhance the oral bioavailability of nutraceuticals in foods due to its inhibitory activity on drug metabolizing enzymes such as cytochrome P450 and p-glycoprotein in the gastrointestinal mucosa. This decreases the first-pass metabolism of nutraceuticals thus increasing their levels in the systemic circulation. Numerous studies in both animals and humans have validated the efficacy of piperine in boosting nutraceutical bioavailability. However, most of these studies utilized highly purified sources of both piperine and nutraceuticals, and therefore do not provide direct evidence on the ability of black pepper (used as a spice) to enhance the bioavailability of nutraceuticals in real foods.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 year old healthy adults

Exclusion Criteria:

* those who are <18 or >30 years old, have a BMI of <20 or >29 kg/m2, have a weight change >4.5 kg (9.91 pounds) in the past 3 months, exceed exercise activities of a recreational level over the past 3 months, have any diseases, especially intestinal disorders including lipid malabsorption or lactose intolerance, had abnormal liver or kidney function tests.
* Those who smoke, consume more than two alcoholic drinks per day, use medication affecting lipid profiles or dietary supplements affecting plasma cholesterol (e.g., Benocol or fiber supplements) will also be excluded.
* Additionally, this study excludes menopausal women, those using hormone-based contraceptives, those with abnormal menstrual cycles, and those who are pregnant, lactating or planning to become pregnant.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Determine the level of carotenoids in blood | 12-16 weeks
  Utilize HPLC to quantify blood levels of carotenoids in subjects consumed test articles

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Applied Life Sciences, Amherst, Massachusetts, United States